CLINICAL TRIAL: NCT00245856
Title: Treatment of Upper Extremity Deep-Vein Thrombosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Suman Rathbun, Professor of Medicine, University of Oklahoma
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10206; ORA-20020622 (Other: University of Oklahoma Office of Research Administration)
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Results first posted 2013-02-04 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Deep-Vein Thrombosis
Keywords: Upper Extremity Deep-Vein Thrombosis; DVT; Fragmin; Deep-Vein Thrombosis; Thrombosis
MeSH Terms: conditions — Venous Thrombosis; Upper Extremity Deep Vein Thrombosis; Thrombosis | interventions — Dalteparin; Warfarin

ARMS (1):
- Treatment of Upper Extremity DVT (Experimental): Participants received dalterparin followed by warfarin or received dalterparin monotherapy for the treatment of upper extremity DVT
  Interventions: Drug: Dalteparin sodium injection; Drug: Warfarin

INTERVENTIONS:
Drug: Dalteparin sodium injection — 200units/kg subcutaneous daily for one month, followed by 150units/kg subcutaneous daily for two additional months or 200 units/kg subcutaneously daily for 5 days followed by warfarin.
  Other Names: Fragmin
Drug: Warfarin — Titrated to INR 2-3 through study month 3

SUMMARY:
The purpose of this study is to document the long-term outcome or prognosis of patients diagnosed with upper extremity deep-vein thrombosis who are treated with Fragmin (dalteparin sodium injection) for three months.

DETAILED DESCRIPTION:
Upper extremity deep-vein thrombosis (DVT) is an increasingly common clinical problem and has been found to cause important pulmonary embolism in up to 36% of cases including fatal embolism. The major risk factor for development of DVT is presence of a central venous catheter in which up to 30% of patients may develop venous thrombosis. Peripherally inserted central catheters or (PICC) lines have been more frequently used in order to avoid the morbidity of central venous catheter insertion. There is little data on the incidence of DVT with these catheters, or effective treatment regimen.

The purpose of this study is to document the long-term outcome or prognosis of patients diagnosed with upper extremity deep-vein thrombosis who are treated with Fragmin (dalteparin sodium injection) for three months. About 100 patients will be enrolled in this study at the University of Oklahoma.

All patients with upper extremity DVT will be screened. Each will have a complete baseline and risk factor assessment.

All patients will receive active study drug for a period of 3 months with reassessment of upper extremity DVT by ultrasound.

All patients will participate for a period of 12 months with follow up visits at 5-7 day, and 1, 3, 6, 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed upper extremity DVT diagnosed by ultrasound imaging or venogram

Exclusion Criteria:

* Active, clinically significant bleeding
* Known hypersensitivity to heparin or low-molecular weight heparin
* Currently pregnant or less than 1 week post-partum
* Acquired bleeding diathesis
* Known inherited bleeding disorder
* Renal failure
* Extremes of weight
* Poor performance status
* Unable to return for repeat diagnostic testing or follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2002-09; Primary Completion 2009-03 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suman W. Rathbun, M.D., Principal Investigator — University of Oklahoma Health Science Center, Dept of Medicine/CardioVascular section
Locations (2):
- United States (2):
  - Department of Veterans Affairs Medical Center, Oklahoma City, Oklahoma
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period November 2002 to December 2008 OUHSC hospital and clinics: OU Medical Center and VA Medical Center
Pre-assignment Details: Consecutive patients, both inpatient and outpatient, who had objectively confirmed upper extremity DVT found on standardized comprehensive duplex imaging or venogram. Ineligibility : predefined ineligibility criteria including high risk of bleeding.
Groups:
- Dalteparin + Warfarin: 200 units per kg with transition Warfarin titrated to INR 2-3
  This arm was completed and new treatment regimen was substituted for the remainder of the study.
- Dalteparin Only: 200 units/kg for one month At month one, dosage reduction based on weight
Period: Period One
Arm/Group | Dalteparin + Warfarin | Dalteparin Only
Started | 28 | 0
Completed | 28 | 0
Not Completed | 0 | 0
Period: Period Two
Arm/Group | Dalteparin + Warfarin | Dalteparin Only
Started | 0 | 39
Completed | 0 | 38
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All DVT Treated Patients: Participants received dalteparin 200units/kg followed by warfarin or dalteparin only for 3 months
Arm/Group | All DVT Treated Patients
Number analyzed (Participants) | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 56
  >=65 years | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 52 (30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 67

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Died at 3 Months
Time Frame: 3 months
Population: All DVT treated patients analyzed together
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All DVT Treated Patients
Number analyzed (Participants) | 66
percentage of participants
  All cause mortality | 8 [3 to 17]
  Deaths attributed to DVT/PE | 0 [NA to NA] — This confidence interval was not calculated

2. Primary Outcome: New Venous Thromboembolism at 3 Months
Description: New DVT or PE at 3 months confirmed by diagnostic testing
Time Frame: 3 months
Population: All DVT treated patients analyzed together
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Dalteparin + Warfarin or Dalteparin Alone: Patients with arm DVT who received either 3 months of dalteparin + warfarin (INR 2-3) or Dalteparin alone
Arm/Group | Dalteparin + Warfarin or Dalteparin Alone
Number analyzed (Participants) | 67
participants | 0 [0 to 5]

3. Secondary Outcome: Bleeding Events
Description: Total major bleeding rate
Time Frame: 3 months
Population: All DVT treated patients analyzed together
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Dalteparin + Warfarin/Dalteparin Alone: Major bleeding rates
Arm/Group | Dalteparin + Warfarin/Dalteparin Alone
Number analyzed (Participants) | 66
participants | 1 [0 to 8]

ADVERSE EVENTS:
Arm/Group | Dalteparin + Warfarin | Dalteparin Only
Serious Adverse Events (participants affected / at risk) | 1/28 | 1/39
Other Adverse Events (participants affected / at risk) | 0/28 | 2/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalteparin + Warfarin (N=28) | Dalteparin Only (N=39)
Bleeding (Blood and lymphatic system disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dalteparin + Warfarin (N=28) | Dalteparin Only (N=39)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No